CLINICAL TRIAL: NCT03206554
Title: Local Infiltration Analgesia in Total Knee Arthroplasty: A Randomized, Prospective, Placebo Controlled, Double Blinded Study.
Brief Title: Local Infiltration Analgesia in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Responsible Party: Principal Investigator, Alexandros Makris, Consultant Anaesthesiologist, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 511/25/09/2015
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Total Knee Arthroplasty; Analgesia
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIA (Active Comparator): Local infiltration analgesia
  Interventions: Drug: Ropivacaine
- sham LIA (Sham Comparator): Saline injections
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Ropivacaine — Large volume local anaesthetic intraarticularly
  Arms: LIA
Other: Saline — sham injection
  Arms: sham LIA

SUMMARY:
40 patients ASA I-III, undergoing total knee arthroplasty were randomly assigned, into one of two groups, namely group LIA (n=20), where local infiltration analgesia would be administered intraoperatively; and group sham LIA (n=20), where sham injections of normal saline would be administered. All patients received a standardized multimodal approach, including pregabalin, adductor canal peripheral nervous blockade, spinal anaesthesia, paracetamol, and PCA with morphine. Morphine consumption during the first 24 hours postoperatively was measured and additionally the investigators recorded: Time of morphine first dose administration, NRS scores in static and dynamic conditions in 6 hours, 12 hours, 18 hours and 24 hours postoperatively, complications, patient satisfaction and duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to American Society of Anesthesiologists (ASA) I-III
* Patients scheduled for total knee arthroplasty

Exclusion Criteria:

* Contraindication for central and/or peripheral nervous blockade
* Reoperation on previous total knee arthroplasty
* History of allergic or other adverse reactions on the agents used in the study
* Chronic opioid or gabapentinoid use
* Serious psychiatric, mental and cognitive disorders
* Language barrier
* Difficulty in understanding or using a patient controlled analgesia device

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours

SECONDARY OUTCOMES:
NRS scores | 24 hours
Complications | 24 hours
Patient satisfaction | 24 hours
  Patients asked whether they would choose the same anaesthetic management in a futue operaton: Yes / No
Duration of hospitalization | 1 month
  Number of days patients remain in the hospital postoperatively

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tziona D, Papaioannou M, Mela A, Potamianou S, Makris A. Local infiltration analgesia combined with a standardized multimodal approach including an adductor canal block in total knee arthroplasty: a prospective randomized, placebo-controlled, double-blinded clinical trial. J Anesth. 2018 Jun;32(3):326-332. doi: 10.1007/s00540-018-2476-x. Epub 2018 Mar 5. PMID 29508066